CLINICAL TRIAL: NCT05306795
Title: Development, Application, and Validation of a Comprehensive Classification Automation System for Allograft Precision Diagnostics in Adult and Pediatric Kidney Transplant Biopsies
Brief Title: Development and Validation of a Comprehensive Classification Automation System for Kidney Allograft Biopsies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Principal Investigator, Professor Alexandre Loupy, Director, Paris Translational Research Center for Organ Transplantation
Other Study IDs: Banff_Automation
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Kidney Transplant Rejection; Pathology
Keywords: Banff classification; Kidney transplantation; Precision diagnostic; Automation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: Observational prospective cohort of kidney transplant allograft biopsies

SUMMARY:
Since 1991, the Banff classification has been the gold standard for defining antibody-mediated rejection (AMR) and T-cell mediated rejection (TCMR), thereby guiding the treatment and management of transplant recipients. Starting from a pure histological approach, the classification has moved over the past three decades towards an integrated precision diagnosis system, which encompasses other expertise, such as immunology, immunogenetic, other basic sciences, biostatistics, data science, and artificial intelligence The counterpart of this constant refinement is that Banff rules are becoming complex to follow, with numerous possible scenarios leading to a high degree of inter-observer variability and misclassifications, which may lead to therapeutic consequences.

The aims of this study are:

1. To integrate and decode all Banff rules and develop a computer-based application - the Banff Automation System - which provides automated and reproducible diagnoses
2. To validate the ability of the Banff Automation System to reclassify rejection diagnoses in multicenter cohort studies and clinical trials.

DETAILED DESCRIPTION:
Despite considerable advances in the development of effective immunosuppressive therapies, allograft rejection remains the main cause of graft loss after kidney transplantation. Since 1991, the Banff classification has been the gold standard for defining antibody-mediated rejection (AMR) and T-cell mediated rejection (TCMR), thereby guiding the treatment and management of transplant recipients. Starting from a pure histological approach, the classification has moved over the past three decades towards an integrated precision diagnosis system, which encompasses other expertise, such as immunology, immunogenetic, other basic sciences, biostatistics, data science, and artificial intelligence The counterpart of this constant refinement is that Banff rules are becoming complex to follow, with numerous possible scenarios leading to a high degree of inter-observer variability and misclassifications, which may lead to therapeutic consequences. Hence, international transplant societies and regulatory agencies urgently appealed for a more comprehensible and reproducible classification, required for decision-making process and reliable surrogate endpoints, to further improve patients care and drug development.

The aims of this study are:

1. To integrate and decode all Banff rules and develop a computer-based application - the Banff Automation System - which provides automated and reproducible diagnoses
2. To validate the ability of the Banff Automation System to reclassify rejection diagnoses in multicenter cohort studies and clinical trials.

Based on the results, the investigators will provide a comprehensive, user-friendly, and open-access online application which might improve reproducibility and precision of biopsies' diagnoses, thereby reducing misclassifications, and path the way to standardize histology-based endpoints in observational studies and clinical trials, and post-transplant diagnostic and therapeutic's management of kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* At least one kidney transplant biopsy performed, assessed with the Banff classification

Exclusion Criteria:

* Inadequate biopsy according to the Banff classification (number of glomeruli inferior less than seven)
* Missing data for Banff lesion scores
* Missing data for donor-specific antibody status
* Missing data for C4d (degradation product of the classic complement pathway) staining

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients of all sexes recruited in observational studies performed in Europe and United States, with at least one kidney biopsy performed with all the relevant data to provide a reliable diagnosis according to the Banff classification (i.e., adequate biopsies without missing data for Banff lesion scores, donor-specific antibody status, and C4d staining).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Rejection-related diagnoses reclassified by the computer-based tool | 1 day (At time of a kidney allograft biopsy)
  Proportion of rejection-related diagnoses reclassified by the computer-based tool

SECONDARY OUTCOMES:
Graft survival | 24 months post-kidney allograft biopsy
  Comparison of graft survival after diagnosis by the computer-based tool

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, MD, PhD, Study Director — Paris Translational Centre for Organ Transplantation
Locations (1):
- Paris Translational Centre for Organ Transplantation, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided
The data analyzed during the current study are available from the Principal investigator on reasonable request including standards for General Data Protection Regulation and Institutional Review Board approval.

REFERENCES:
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180
- [Background] Haas M, Loupy A, Lefaucheur C, Roufosse C, Glotz D, Seron D, Nankivell BJ, Halloran PF, Colvin RB, Akalin E, Alachkar N, Bagnasco S, Bouatou Y, Becker JU, Cornell LD, Duong van Huyen JP, Gibson IW, Kraus ES, Mannon RB, Naesens M, Nickeleit V, Nickerson P, Segev DL, Singh HK, Stegall M, Randhawa P, Racusen L, Solez K, Mengel M. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 2018 Feb;18(2):293-307. doi: 10.1111/ajt.14625. Epub 2018 Jan 21. PMID 29243394
- [Background] Loupy A, Haas M, Solez K, Racusen L, Glotz D, Seron D, Nankivell BJ, Colvin RB, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell L, Drachenberg C, Dragun D, de Kort H, Gibson IW, Kraus ES, Lefaucheur C, Legendre C, Liapis H, Muthukumar T, Nickeleit V, Orandi B, Park W, Rabant M, Randhawa P, Reed EF, Roufosse C, Seshan SV, Sis B, Singh HK, Schinstock C, Tambur A, Zeevi A, Mengel M. The Banff 2015 Kidney Meeting Report: Current Challenges in Rejection Classification and Prospects for Adopting Molecular Pathology. Am J Transplant. 2017 Jan;17(1):28-41. doi: 10.1111/ajt.14107. PMID 27862883
- [Background] Mengel M, Loupy A, Haas M, Roufosse C, Naesens M, Akalin E, Clahsen-van Groningen MC, Dagobert J, Demetris AJ, Duong van Huyen JP, Gueguen J, Issa F, Robin B, Rosales I, Von der Thusen JH, Sanchez-Fueyo A, Smith RN, Wood K, Adam B, Colvin RB. Banff 2019 Meeting Report: Molecular diagnostics in solid organ transplantation-Consensus for the Banff Human Organ Transplant (B-HOT) gene panel and open source multicenter validation. Am J Transplant. 2020 Sep;20(9):2305-2317. doi: 10.1111/ajt.16059. Epub 2020 Jun 27. PMID 32428337
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190
- [Background] Mengel M, Sis B, Haas M, Colvin RB, Halloran PF, Racusen LC, Solez K, Cendales L, Demetris AJ, Drachenberg CB, Farver CF, Rodriguez ER, Wallace WD, Glotz D; Banff meeting report writing committee. Banff 2011 Meeting report: new concepts in antibody-mediated rejection. Am J Transplant. 2012 Mar;12(3):563-70. doi: 10.1111/j.1600-6143.2011.03926.x. Epub 2012 Feb 2. PMID 22300494
- [Background] Sis B, Mengel M, Haas M, Colvin RB, Halloran PF, Racusen LC, Solez K, Baldwin WM 3rd, Bracamonte ER, Broecker V, Cosio F, Demetris AJ, Drachenberg C, Einecke G, Gloor J, Glotz D, Kraus E, Legendre C, Liapis H, Mannon RB, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Rodriguez ER, Seron D, Seshan S, Suthanthiran M, Wasowska BA, Zachary A, Zeevi A. Banff '09 meeting report: antibody mediated graft deterioration and implementation of Banff working groups. Am J Transplant. 2010 Mar;10(3):464-71. doi: 10.1111/j.1600-6143.2009.02987.x. Epub 2010 Jan 29. PMID 20121738
- [Background] Solez K, Colvin RB, Racusen LC, Sis B, Halloran PF, Birk PE, Campbell PM, Cascalho M, Collins AB, Demetris AJ, Drachenberg CB, Gibson IW, Grimm PC, Haas M, Lerut E, Liapis H, Mannon RB, Marcus PB, Mengel M, Mihatsch MJ, Nankivell BJ, Nickeleit V, Papadimitriou JC, Platt JL, Randhawa P, Roberts I, Salinas-Madriga L, Salomon DR, Seron D, Sheaff M, Weening JJ. Banff '05 Meeting Report: differential diagnosis of chronic allograft injury and elimination of chronic allograft nephropathy ('CAN'). Am J Transplant. 2007 Mar;7(3):518-26. doi: 10.1111/j.1600-6143.2006.01688.x. PMID 17352710
- [Background] Racusen LC, Halloran PF, Solez K. Banff 2003 meeting report: new diagnostic insights and standards. Am J Transplant. 2004 Oct;4(10):1562-6. doi: 10.1111/j.1600-6143.2004.00585.x. PMID 15367210
- [Background] Solez K, Axelsen RA, Benediktsson H, Burdick JF, Cohen AH, Colvin RB, Croker BP, Droz D, Dunnill MS, Halloran PF, et al. International standardization of criteria for the histologic diagnosis of renal allograft rejection: the Banff working classification of kidney transplant pathology. Kidney Int. 1993 Aug;44(2):411-22. doi: 10.1038/ki.1993.259. PMID 8377384
- [Background] Loupy A, Mengel M, Haas M. Thirty years of the International Banff Classification for Allograft Pathology: the past, present, and future of kidney transplant diagnostics. Kidney Int. 2022 Apr;101(4):678-691. doi: 10.1016/j.kint.2021.11.028. Epub 2021 Dec 17. PMID 34922989
- [Background] Solez K, Colvin RB, Racusen LC, Haas M, Sis B, Mengel M, Halloran PF, Baldwin W, Banfi G, Collins AB, Cosio F, David DS, Drachenberg C, Einecke G, Fogo AB, Gibson IW, Glotz D, Iskandar SS, Kraus E, Lerut E, Mannon RB, Mihatsch M, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Roberts I, Seron D, Smith RN, Valente M. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant. 2008 Apr;8(4):753-60. doi: 10.1111/j.1600-6143.2008.02159.x. Epub 2008 Feb 19. PMID 18294345
- [Background] Racusen LC, Solez K, Colvin RB, Bonsib SM, Castro MC, Cavallo T, Croker BP, Demetris AJ, Drachenberg CB, Fogo AB, Furness P, Gaber LW, Gibson IW, Glotz D, Goldberg JC, Grande J, Halloran PF, Hansen HE, Hartley B, Hayry PJ, Hill CM, Hoffman EO, Hunsicker LG, Lindblad AS, Yamaguchi Y, et al. The Banff 97 working classification of renal allograft pathology. Kidney Int. 1999 Feb;55(2):713-23. doi: 10.1046/j.1523-1755.1999.00299.x. PMID 9987096
- [Background] Racusen LC, Colvin RB, Solez K, Mihatsch MJ, Halloran PF, Campbell PM, Cecka MJ, Cosyns JP, Demetris AJ, Fishbein MC, Fogo A, Furness P, Gibson IW, Glotz D, Hayry P, Hunsickern L, Kashgarian M, Kerman R, Magil AJ, Montgomery R, Morozumi K, Nickeleit V, Randhawa P, Regele H, Seron D, Seshan S, Sund S, Trpkov K. Antibody-mediated rejection criteria - an addition to the Banff 97 classification of renal allograft rejection. Am J Transplant. 2003 Jun;3(6):708-14. doi: 10.1034/j.1600-6143.2003.00072.x. PMID 12780562
- [Background] Solez K, Hansen HE, Kornerup HJ, Madsen S, Sorensen AW, Pedersen EB, Marcussen N, Benediktsson H, Racusen LC, Olsen S. Clinical validation and reproducibility of the Banff schema for renal allograft pathology. Transplant Proc. 1995 Feb;27(1):1009-11. No abstract available. PMID 7878779
- [Background] Solez K, Benediktsson H, Cavallo T, Croker B, Demetris AJ, Drachenberg C, Emancipator S, Furness PN, Gaber LW, Gibson IW, Gough J, Gupta R, Halloran P, Hayry P, Kashgarian M, Marcussen N, Massy ZA, Mihatsch MJ, Morozumi K, Noronha I, Olsen S, Papadimitriou J, Paul LC, Picken M, Racusen LC, Ramos EL, Randhawa P, Rayner DC, Rush D, Sanfilippo F, Taskinen E, Trpkov K, Truong L, Yamaguchi Y, Yilmaz S. Report of the Third Banff Conference on Allograft Pathology (July 20-24, 1995) on classification and lesion scoring in renal allograft pathology. Transplant Proc. 1996 Feb;28(1):441-4. No abstract available. PMID 8644308
- [Derived] Yoo D, Goutaudier V, Divard G, Gueguen J, Astor BC, Aubert O, Raynaud M, Demir Z, Hogan J, Weng P, Smith J, Garro R, Warady BA, Zahr RS, Sablik M, Twombley K, Couzi L, Berney T, Boyer O, Duong-Van-Huyen JP, Giral M, Alsadi A, Gourraud PA, Morelon E, Le Quintrec M, Brouard S, Legendre C, Anglicheau D, Villard J, Zhong W, Kamar N, Bestard O, Djamali A, Budde K, Haas M, Lefaucheur C, Rabant M, Loupy A. An automated histological classification system for precision diagnostics of kidney allografts. Nat Med. 2023 May;29(5):1211-1220. doi: 10.1038/s41591-023-02323-6. Epub 2023 May 4. PMID 37142762